CLINICAL TRIAL: NCT05570123
Title: Effect and Tolerance of Standardized Exclusive Dry Extracts of Curcuma Longa (CURTIL03) and of Boswellia Serrata (BOSTIL01) in Support of Standard Treatments Among People With Hand Joint Discomfort and Dysfunction: a Multicenter Hospital Setting, Randomized, Blinded, Placebo-controlled Clinical Study.
Brief Title: Effect and Tolerance of Standardized Exclusive Dry Extracts of Curcuma Longa and of Boswellia Serrata Among People With Hand Joint Discomfort and Dysfunction
Acronym: FLEXOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tilman S.A. (Industry)
Collaborators: Artialis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FLEXOA
Record Dates: First submitted 2022-10-05; First posted 2022-10-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-01

CONDITIONS: Hand Joint Discomfort; Hand Joint Dysfunction
Keywords: Hand joint pain; Curcuma; Boswellia; Flexofytol Forte

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Flexofytol Forte (Experimental)
  Interventions: Dietary Supplement: Flexofytol Forte

INTERVENTIONS:
Dietary Supplement: Flexofytol Forte — standardized exclusive dry extracts of Curcuma longa and Boswellia serrata. 2 tablets a day, one in the morning, one in the evening
  Arms: Flexofytol Forte
Dietary Supplement: Placebo — 2 tablets a day, one in the morning, one in the evening
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the effect and tolerance of standardized exclusive dry extracts of Curcuma longa (CURTIL03) and of Boswellia serrata (BOSTIL01) among people with hand joint discomfort and dysfunction.

The study is prospective, randomized, double-blinded, placebo-controlled with 2 parallel-groups in 200 participants. The study is multicentric and will be done by 11 investigators located in Belgium including rheumatologists, sports and rehabilitation physicians, physical therapists, or any hand articular disease specialists.

DETAILED DESCRIPTION:
200 adult subjects suffering from significant hand joint discomfort will be randomized per site in 2 parallel groups (100 subjects per group).

Each patient will be enrolled in the study for 3 months including 3 visits: Inclusion/Baseline visit (V0), follow-up visits after 1 month (V1) and 3 months (V2).

A-PRIMARY OBJECTIVE Evaluate the effect of the association of standardized exclusive dry extracts of Curcuma longa CURTIL03 and Boswellia serrata BOSTIL01 versus placebo on the fingers pain after 3 months supplementation.

B-SECONDARY OBJECTIVES

Evaluate:

* finger pain on both hands at 1 month (mean and AUC) and 3 months (AUC)
* Functional disability at any timepoint (self-administrate questionnaire)
* Participant Global Assessment (PGA) at any timepoint
* To evaluate Minimum Clinically Important Improvement (MCII)
* To calculate Participant Acceptable important Symptom State (PASS)
* Consumption of rescue treatment (Paracetamol and oral NSAIDS) for hand pain at any timepoint
* Tender and swollen joints at any timepoint
* Grip strength at any timepoint
* Quality of life (e.g. including mood, sleep, disability) at any timepoint
* Tolerance to the product at 1 and 3 months
* Compliance to the product at 1 and 3 months
* Responder to supplementation at 1 and 3 months

EXPLORATIVE OBJECTIVES

• Evaluate the blood level of cartilage catabolism and inflammatory biomarkers before and after 3 months of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≤ 35 kg/m2
* Subjects that fulfil the following American College of Rheumatology (ACR) clinical criteria :

  * Hand pain, aching, or stiffness AND
  * 3 or 4 of the following features:

    * Hard tissue enlargement of 2 or more of 10 selected joints,
    * Hard tissue enlargement of 2 or more Distal interphalangeal (DIP) joints,
    * Fewer than three swollen metacarpophalangeal (MCP) joints,
    * Deformity of at least 1 of 10 selected hand joints.

The 10 selected joints are the second and third Distal Interphalangeal joint (DIP), the second and third Proximal Interphalangeal joints (PIP), and the first carpometacarpal (CMC) joints of both hands.

* Pain in hands at least half of the days in the previous month and for at least 48 h prior to the inclusion/baseline visit.
* Finger pain score of 40-80 mm on a 100 mm Visual Analog Scale (VAS) on at least one hand over the last 24 hours. Subjects should respect a 24-hours wash-out period of authorized analgesic/anti-inflammatory medications (Paracetamol/oral NSAIDs) before the visit.
* Willing to use only Paracetamol and oral NSAIDS as rescue treatment to manage hand pain during the study. Others analgesics and anti-inflammatory medication (oral and topic) are not allowed during the study and a wash out period of 5 half-life depending of the molecule should be respected before study entry.
* Able to follow the instructions of the study
* Having signed an informed consent

Exclusion Criteria:

Subjects that meet AT LEAST one of the following criteria will be excluded:

Related to hand

* Subjects with discomfort uniquely of thumb joints.
* Other rheumatic diseases such gout, rheumatoid arthritis, psoriatic arthritis, to name a few) should be excluded.
* Concurrent articular diseases or hand/upper limb disorders interfering with the evaluation of hand pain such as but not limited to inflammatory arthritis, connective tissue disorder, chronic pain or alternative clinical diagnosis such as tenosynovitis or carpal tunnel syndrome, such as poly-articular chondrocalcinosis, thoracic outlet syndrome, carpal tunnel, Guyon's canal syndrome, cubital tunnel syndrome, diabetic neuropathy or cheiroarthropathy, palmar tenosynovitis, trigger finger, fibromyalgia, pain syndrome (Complex Regional Pain Syndrome or algoneurodystrophy) diagnosed within past 6 months (left to Principal Investigator (PI) discretion).
* Major injury in hand joint(s) and tendons within past 6 months (left to PI discretion).

Related to treatments

* Analgesics and anti-inflammatory medications (oral and topic) other than Paracetamol and oral NSAIDS at inclusion except if a wash-out period is respected.
* Intra-articular corticosteroids in past 3 months in any joint.
* Intra-articular Hyaluronic Acid in any hand/finger joint within past 6 months.
* Intra-articular platelet-rich plasma in any hand/finger joint within past 6 months.
* Use of Slow-acting drugs for OA (SYSADOA) and/or dietary supplements in the last 3 months (e.g. chondroitin sulfate, diacerein, soy and avocado unsaponifiables, collagen, hyaluronic acid, oxaceprol, copper granions, glucosamine, phytotherapy for joints pain and dysfunction, homeopathy for joints pain and dysfunction, dietary supplements based on curcumin and/or Boswellic acids)
* Oral corticotherapy ≥ 5mg/day (in Prednisolone equivalent) in the last 3 months
* Allergy or contra-indication to the studied product or any ingredient present in this product or in placebo. Attention to medication interaction, see section on prohibited treatments
* Intolerance to Paracetamol and NSAIDS (rescue treatments during the study)
* Anticoagulant (coumarin compound) and heparin. New generation anticoagulants are authorized
* Anticipated need for any joint discomfort including OA treatments forbidden during the study
* Hand surgery or fracture within the last 6 months, or hand surgery planned within the next 3 months
* Physiotherapy for hand pain and dysfunction in the past month.

Related to associated diseases

* Severe and uncontrolled diseases (such as peptic ulcer, renal impairment, hepatic dysfunction, hematologic disease, cancer within 5 years (except treated Basal Cell Carcinoma, BCC), HIV, etc.)
* Participants who cannot swallow tablets because of the size of the tablets that cannot be cut or disintegrated.
* Any other significant or uncontrolled disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study (as disease with widespread pain)

Related to subjects

* Close collaborators to the investigational team, the study coordinator (ARTIALIS) or the Sponsor (TILMAN)
* Having participated or currently participating to a clinical trial in the last 3 months
* Vegan people (the product contains bovine gelatin)
* Under guardianship or judicial protection
* Pregnancy, breastfeeding, planned conception
* Women of childbearing age without contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to 3 months of mean finger pain during the last 24 hours | 3 months (between V0 and V2 visits)
  0 -100 mm Visual Analog Scale (VAS)-From 0 (No pain) to 100 (maximal pain)

SECONDARY OUTCOMES:
Changes from baseline to 1 month of Mean finger pain evaluated in both hands during the last 24 hours | 1 month (between V0 and V1 visits)
  0 -100 mm Visual Analog Scale (VAS)-From 0 (No pain) to 100 (maximal pain)
Changes from baseline to 1 month of AUC finger pain intensity evaluated in both hands during the last 24 hours | 1 month (between V0 and V1 visits)
  0 -100 mm Visual Analog Scale (VAS)-From 0 (No pain) to 100 (maximal pain)
Changes from baseline to 1 month of functional disability | 1 month (between V0 and V1 visits)
  Functional Index For Hand Osteoarthritis (FIHOA) self-reported questionnaire-from 0 (no functional impairment) to 30 points (maximal impairment)
Changes from baseline to 1 month of PGA | 1 month (between V0 and V1 visits)
  0 -100 mm Visual Analog Scale (VAS)-From 0 (No impact) to 100 (maximal impact)
Changes from baseline to 1 month of Minimum Clinically Important improvement (MCHII) | 1 month (between V0 and V1 visits)
  Calculated on Visual Analog Scale (finger pain)-absolute change of 15 mm or relative change of 20%
Changes from baseline to 1 month of Participant Acceptable important Symptom State (PASS) | 1 month (between V0 and V1 visits)
  Calculated on Visual Analog Scale (finger pain)- < 40 mm
Changes from baseline to 1 month of tender and /or swollen joints counts | 1 month (between V0 and V1 visits)
Changes from baseline to 1 month of Grip strength of both hands | 1 month (between V0 and V1 visits)
  measured by dynamometer-0 to 90 Kilograms-increased strength defines an improvement in hand function
Changes from baseline to 1 month of quality of life | 1 month (between V0 and V1 visits)
  using Short Form (SF)-36 questionnaire-0 to 100 range-high score defines a more favorable health state
Changes from baseline to 1 month of consumption of paracetamol and oral NSAIDS | 1 month (between V0 and V1 visits)
  recording via a diary
Changes from baseline to 3 months of functional disability | 3 months (between V0 and V3 visits)
  FIHOA self-reported questionnaire-from 0 (no functional impairment) to 30 points (maximal impairment)
Changes from baseline to 3 months of PGA | 3 months (between V0 and V3 visits)
  0 -100 mm Visual Analog Scale (VAS)-From 0 (No impact) to 100 (maximal impact)
Changes from baseline to 3 months of Minimum Clinically Important improvement (MCHII) | 3 months (between V0 and V3 visits)
  Calculated on Visual Analog Scale (finger pain)-absolute change of 15 mm or relative change of 20%
Changes from baseline to 3 months of Participant Acceptable important Symptom State | 3 months (between V0 and V3 visits)
  Calculated on Visual Analog Scale (finger pain)- < 40 mm
Changes from baseline to 3 months of tender and /or swollen joints counts | 3 months (between V0 and V3 visits)
Changes from baseline to 3 months of Grip strength of both hands | 3 months (between V0 and V3 visits)
  measured by dynamometer-0 to 90 Kilograms-increased strength defines an improvement in hand function
Changes from baseline to 3 months of quality of life | 3 months (between V0 and V3 visits)
  using SF-36 questionnaire-0 to 100 range-high score defines a more favorable health state
Changes from baseline to 3 months of consumption of paracetamol and oral NSAIDS | 3 months (between V0 and V3 visits)
  recording via a diary
Tolerance | 3 months (between V0 and V3 visits)
  Record of adverse and Serious Adverse Events (AE; SAE) and drop-outs
Compliance | 3 months (between V0 and V3 visits)
  Tablet count by the investigator
Fulfillment of Osteoarthritis Research Society International (OARSI) responder criteria from OMERACT(Outcome Measures in Rheumatoid Arthritis Clinical Trials)-OARSI initiative | 3 months (between V0 and V3 visits)

OTHER OUTCOMES:
Change from baseline to 3 months in blood levels of cartilage metabolism and inflammatory biomarkers | 3 months (between V0 and V3 visits)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Wittoek (National coordinator), Pr, MD, Principal Investigator — UZ Gent
Locations (1):
- UZ Gent (national coordinating site), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No